CLINICAL TRIAL: NCT03487133
Title: A Prospective, Multi-center, Open-label, Single-arm, Phase II Study of Bortezomib/Dexamethasone Therapy in Patients With Relapsed and/or Refractory Cutaneous T-cell Lymphoma
Brief Title: Bortezomib/Dexamethasone Therapy in Patients With Relapsed and/or Refractory Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-104
Record Dates: First submitted 2018-01-18; First posted 2018-04-03 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Relapsed and/or Refractory Cutaneous T-cell Lymphoma
MeSH Terms: interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bortezomib/dexamethasone (Experimental): Subjects who have been diagnosed with stable lesions more than 4 cycles of induction therapy (Induction Therapy Part I) will receive additional induction therapy 4 cycles (Induction Therapy Part II) Patients who have been diagnosed with a stable disease response after a total of eight cycles of induction therapy receive up to one year of maintenance therapy.
  Interventions: Drug: bortezomib/dexamethasone

INTERVENTIONS:
Drug: bortezomib/dexamethasone — Induction therapy ->1cycle=28 days 1,2,3week : bortezomib 1.6 mg/m2 SC(subcutaneous), dexamethasone 40mg IV 4week : none maintenance therapy ->1cycle=28 days
  1week : bortezomib 1.6 mg/m2 SC(subcutaneous), dexamethasone 40mg IV 2,3,4week : none

SUMMARY:
the efficacy and safety of bortezomib / dexamethasone combination therapy in patients with relapsed or refractory T-cell lymphoma who have failed one or more treatments.

* primary purpose

  1. Overall response rate
* secondary purpose

  1. Progression-free survival and overall survival
  2. Disease stabilization ratio
  3. Duration of reaction
  4. Safety Profile
  5. Experiments on response prediction / immunological markers

DETAILED DESCRIPTION:
In a Phase II study in patients with previous T-cell lymphoma, bortezomib was administered at a dose of 1.6 mg / m 2 on Day 1 and Day 8, and combined with CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone) chemotherapy . The 1.6 mg / m2 dose of bortezomib was obtained through phase 1 studies, and the Phase II study included five patients with skin T-cell lymphoma, with an overall response rate of 87%. In addition, there was no significant increase in toxicity when bortezomib was administered at 1.6 mg / m2 every week. The fact that there was no increase in toxicity in combination with a drug commonly used to induce peripheral neuropathy, such as vincristine, / m2 suggests the safety of the dosage at 1 week intervals.Therefore, in order to improve the convenience of administration with once-weekly dosing, this study combined 1.6 mg / m2 every week for 1 week, 2 weeks, and 3 weeks in a 4-week cycle, The dose was determined by a single dose.In addition, it is known that the main dose-limiting toxicity of subcutaneous injection is significantly reduced in peripheral neuropathy, so the route of administration was determined to be via subcutaneous administration (18).Considering that one of the major difficulties in remediation of skin T-cell lymphoma is the short duration of the response after termination of treatment, the subjects who were considered to have a response to the test drug, that is, those who acquired a stable lesion response after 8 cycles of induction therapy The test was designed so that maintenance therapy can be performed up to one year.Even with one year of maintenance therapy, there is no safety concern since the cumulative dose of the test drug is not higher than the cumulative dose currently used as the primary treatment for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed subcutaneous skin T-cell lymphoma based on the WHO(World Health Organization)-EORTC classification (mycosis fungoides, Sezary syndrome,primary cutaneous anaplastic large cell lymphoma,lymphomatoid papulosis,primary cutaneous peripheral T-cell lymphoma, unspecified)
* Male and female patients aged 19-80
* ECOG(Eastern Cooperative Oncology Group performance) 0~2
* Presence of measurable lesion according to ISCL(International Society for Cutaneous Lymphomas)-USCLC(United States Cutaneous Lymphoma Consortium)-EORTC(European Organization of Research and Treatment of Cancer) recommendation
* If one or more of the previous treatments fails or has recurred / progressed
* Proper function status of bone marrow, kidney, liver
* All toxic effects due to previous treatment have been resolved to CTCAE 4.03 version 1 or lower
* For pregnant women, the result of pregnancy test is negative. (The pregnant female patient should have effective contraception during the treatment period and for one month thereafter) (ie, hormonal contraceptive device, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) Men should use effective contraception during the treatment period and for three months thereafter.)
* Patients who are expected to follow and comply with the clinical trial protocol at the discretion of the tester
* Patients who voluntarily agreed to participate in this trial and signed a consent form
* Patients who agreed to donate a sample of peripheral lesions (10 unstained slides) and 3 ml of peripheral blood after baseline and cycle 8

Exclusion Criteria:

* Patients undergoing chemotherapy at the time of clinical trials
* Patients who are undergoing radiotherapy at the time of their participation in the trial or who received radiotherapy within the first 6 months of the trial. However, patients who have additional lesions elsewhere in the main lesion may be eligible for clinical trials if they have completed local radiotherapy as a palliative treatment prior to the administration of the drug, and recovered from the resulting toxicity.
* Patients with symptomatic or uncontrolled angina and congestive heart failure, arrhythmia requiring drug therapy, significant risk of clinically significant myocardial infarction within 6 months prior to participation in this trial
* Patients with stable left ventricular ejection fraction less than the normal lower limit of each organ.
* Adverse Reactions Common Terminology Criteria 4.03 In case of infection in excess of grade 2 according to the standards. Hepatitis B is allowed if there is no active replication (HBV DNA> 20,000 iU / mL associated with ALT(alanine aminotransferase) exceeding twice the normal upper limit).
* If there is active infection, including severe concomitant disease and / or active hepatitis C and human immunodeficiency virus infection
* Patients who received chemotherapy, surgical treatment (permissive for mild surgical treatment) within 4 weeks of the administration of this drug
* History of allogeneic transplantation (including hematopoietic stem cell transplantation)
* Patients with a malignant tumor other than the target disease. However, the following cases are allowed.If you have not received treatment for the tumor for at least 5 years or have no disease,Complete resection of basal cell carcinoma / squamous cell carcinoma or at least 1 year after successful treatment of cervical intraepithelial cancer
* Adverse reactions within 30 days prior to the start of screening Common Grade Criteria 4.03 Severe gastrointestinal bleeding in excess of grade 2
* The occurrence of thrombosis or embolism within 6 months before screening
* Patients with central nervous system involvement.
* Pregnant, lactating, or reproductive women who are not willing to use appropriate contraception during the trial
* Unstable conditions that may impair patient safety and compliance with the test
* Patients with seizure disorders requiring medication
* If you have substance abuse, medical, mental or social illnesses that may interfere with the patient's participation in the clinical trial or the evaluation of clinical trial results
* Patients with a history of hypersensitivity to Drug or Drug component (bortezomib, boron, mannitol, dexamethasone)
* Patients with Acute Diffuse Invasive Pulmonary Disease and Cardiovascular Disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate of tumor | Through study completion, an average of 3 years
  Overall response rate (complete remission, partial remission) according to the ISCL-USCLC-EORTC recommendation evaluated by institutional investigators

SECONDARY OUTCOMES:
progressive-free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 72 months
  the time interval between the first clinical trial dosing date and the first occurring date of tumor progression or death (due to all causes) Duration of response: The time from the first documentation of the objective tumor response to the time of disease progression or death (due to all causes)
Disease stabilization rate | An average of 6 years
  Percentage of subjects who achieved complete remission, partial remission, or stable lesions as a result of tumor response
Duration of response | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 72 months
  The time from the first documentation of the objective tumor response to the time of disease progression or death (due to all causes)

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, Study Chair — 81, Irwon-Ro, Gangnam-Gu, Seoul, Korea 135-710
Locations (1):
- Samsung medical center, Seoul, Gang Nam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] (1) Bradford PT, et al. Blood 2009; 113: 5064 (2) Criscione VD, et al. Arch Dermatol 2007; 143: 854 (3) Willemze R. et al. Blood 2005; 105: 3768 (4) Li JY, et al. Cancer Manag Res 2012; 4: 75 (5) Wilcox RA. Am J Hematol 2016; 91: 152 (6) Querfeld C, et al. Blood 2014; 123: 1159 (7) Kim YH, et al. J Am Acad Dermatol 2010; 63: 975 (8) Yamamoto K, et al. J Clin Oncol 2010; 28: 1591 (9) Bose P, et al. Exp Opin Pharmacother 2014; 15: 2443 (10) Manfé V, et al. PLoS One 2013; 8: e59390 (11) Chang TP, et al. Am J Cancer Res 2013; 3: 433 (12) Chang TP, et al. J Immunol 2015; 194: 1942 (13) Ungewickell A, et al. Nat Genet 2015; 47: 1056 (14) Jagannath S, et al. Br J Haematol 2005; 129: 776 (15) Jagannath S, et al. Br J Haematol 2009; 146: 619 (16) Zinzani PL, et al. J Clin Oncol 2007; 25: 4293 (17) Kim SJ, et al. Eur J Cancer 2012; 48: 3223 (18) Moreau P, et al. Lancet Oncol 2011; 12: 431